CLINICAL TRIAL: NCT07158216
Title: LONG-TERM EFFECT OF TRANSCRANIAL MAGNETIC STIMULATION AND TRANSCRANIAL ELECTRICAL STIMULATION IN PRIMARY PROGRESSIVE APHASIA: RANDOMIZED, DOUBLE-BLIND CLINICAL TRIAL (RECONNECT-PLUS)
Brief Title: Long Term Effect of Brain Stimulation in PPA
Acronym: RECONNECT-PLUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jordi A Matias-Guiu, MD PhD Neurologist, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hospital Clinico San Carlos
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Progressive Aphasia(PPA)
Keywords: Primary progressive aphasia; Frontotemporal dementia; Alzheimer's disease; Brain stimulation; Transcranial Magnetic Stimulation; Transcranial direct current stimulation; Transcranial electrical stimulation
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both outcome assessors and participants will be blinded to the assigned treatment. Only the technicians administering TMS will be aware of the brain stimulation assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- active TMS + active tDCS (Experimental)
  Interventions: Device: TMS; Device: tDCS
- active TMS + sham tDCS (Experimental)
  Interventions: Device: TMS; Device: Sham tDCS
- sham TMS + active tDCS (Experimental)
  Interventions: Device: tDCS; Device: Sham TMS
- sham TMS + sham tDCS (Sham Comparator)
  Interventions: Device: Sham TMS; Device: Sham tDCS

INTERVENTIONS:
Device: TMS — Active TMS + sham tDCS. All patients will receive language therapy immediately after brain stimulation. The period of treatment will be 6 months, comprising 10 consecutive sessions in two weeks (intensive period) followed by once per week (maintenance period of 22 weeks)
  Arms: active TMS + active tDCS; active TMS + sham tDCS
Device: tDCS — sham TMS + active tDCS. All patients will receive language therapy immediately after brain stimulation. The period of treatment will be 6 months, comprising 10 consecutive sessions in two weeks (intensive period) followed by once per week (maintenance period of 22 weeks)
  Arms: active TMS + active tDCS; sham TMS + active tDCS
Device: Sham TMS — Sham TMS. All patients will receive language therapy immediately after brain stimulation. The period of treatment will be 6 months, comprising 10 consecutive sessions in two weeks (intensive period) followed by once per week (maintenance period of 22 weeks)
  Arms: sham TMS + active tDCS; sham TMS + sham tDCS
Device: Sham tDCS — Sham tDCS. All patients will receive language therapy immediately after brain stimulation. The period of treatment will be 6 months, comprising 10 consecutive sessions in two weeks (intensive period) followed by once per week (maintenance period of 22 weeks)
  Arms: active TMS + sham tDCS; sham TMS + sham tDCS

SUMMARY:
The goal of this clinical trial is to investigate the effect of non-invasive brain stimulation techniques in the progression of primary progressive aphasia for 6 months. We will compare three modalities of brain stimulation (TMS, tDCS, TMS+tDCS) against sham stimulation. All patients will receive also language therapy.

DETAILED DESCRIPTION:
Transcranial Magnetic Stimulation will follow an intermitent theta-burst protocol targetting the left dorsolateral prefrontal cortex. Transcranial electrical stimulation will also follow an excitatory protocol over the same region. All brain stimulation procedures will be conducted under neuronavigation. Language therapy will follow the lexical retrieval cascade protocol and will be conducted after each brain stimulation session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPA according to the current consensus criteria supported by neuroimaging (FDG-PET or MRI) (Gorno-Tempini et al., 2011);
* Clinical Dementia Rating scale equal or less than 1;
* The language impairment is the main neurological deficit for the patient.

Exclusion Criteria:

* Patient diagnosed with a condition other than PPA that could cause language impairment;
* History of epilepsy or presence of focal epileptiform pathology on EEG recording; ·Contraindications related to the treatments or procedures to be used (TMS and tDCS), such as ferromagnetic material, pregnancy, or breastfeeding;
* Terminal illness or active malignancy;
* Alcohol or substance abuse within the past year;
* Major psychiatric disorders (schizophrenia, schizoaffective disorders, bipolar disorder, obsessive-compulsive disorder, or personality disorders);
* Absolute inability to communicate (mutism), or poor command of the language that, in the investigator's judgment, would prevent participation in the study;
* Severity of PPA that prevents participation in interventions or assessments at the time of inclusion;
* Participation in another clinical trial within the previous 4 months;
* Chronic use of medications that could affect study outcomes;
* Antiepileptic drugs: allowed if on stable doses for at least 3 months before inclusion. If needed during the study due to seizure occurrence, they may be added;
* Diazepam and derivatives: permitted only if on stable doses for at least 3 months before inclusion. Dose adjustments during the study are allowed;
* Donepezil, Galantamine, Rivastigmine, and Memantine: allowed if on stable doses for at least 3 months before inclusion;
* SSRIs (Selective Serotonin Reuptake Inhibitors): permitted only if on stable doses for at least 3 months prior to inclusion. If necessary during the study, they may be added;
* Medications that may lower the seizure threshold (e.g., tricyclic antidepressants, antipsychotics): allowed if on stable doses for at least 3 months before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mini-Linguistic State Examination | 6 months

SECONDARY OUTCOMES:
Naming of trained words | 6 monhts
  It will be evaluated using a list of 261 words from eight semantic categories (animals, food, objects, places, furniture, clothing, transportation, and body parts)
ACE-III | 6 months
  General cognition
Interview for Deterioration in Daily Living Activities in Dementia (IDDD) | 6 months
  Functional activities
Communicative Effectiveness Index (CETI) | 6 months
  Functional communication questionnaire
CDR(R) plus NACC FTLD-SB | 6 months
  Clinical Dementia Rating
Neuropsychiatric Inventory (NPI) | 6 months
  Neuropsychiatric symptoms
FDG-PET imaging | 6 months
  Regional brain metabolism in a region of interest capturing a large part of the left hemisphere and associated with clinical decline in PPA (Fernandez-Romero et al. 2025)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain